CLINICAL TRIAL: NCT00661700
Title: A Double-blind "Preferred" Vardenafil Dose Study of QoL and Functional Outcomes in Males With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10940; CTX0010/0267/A
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Quality of Life
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10mg Vardenafil for 4 weeks followed by an 8 week titration period when subjects may be titrated up to 20mg Vardenafil or down to 5mg Vardenafil followed by 14 weeks treatment at preferred dose.
  Arms: Arm 1
Drug: Placebo — 10mg placebo for 4 weeks followed by an 8 week titration period when subjects may be titrated up to 20mg placebo or down to 5mg placebo followed by 14 weeks placebo at preferred dose
  Arms: Arm 2

SUMMARY:
To find out more information on how treating impotence with vardenafil in comparison to placebo affects the quality of life (QoL) of men and their partners. Subjects will receive 10mg vardenafil or placebo for 4 weeks followed by an 8 week period when the dose of vardenafil may be reduced to 5mg or increased to 20mg. Subjects will then receive their 'preferred' dose for 14 weeks. During this time Quality of Life Measures will be collected via questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Males with erectile dysfunction for more than six months according to the NIH Consensus Statement (the inability to achieve or maintain penile erection sufficient for satisfactory sexual performance)

  * Stable, heterosexual relationship for more than six months
  * Documented written Informed Consent, from both the patient and his partner, after receiving adequate previous information and prior to any study specific procedures.
* An ED-EQoL score < or = 15.- An IIEF score < or = 25.

Exclusion Criteria:

* Presence of penile anatomical abnormalities (eg. penile fibrosis or Peyronie's disease) that would significantly impair erectile function.
* History of radical prostatectomy. - Retinitis pigmentosa.
* History of positive test for Hepatitis B surface antigen (HbsAg) or Hepatitis C.- Unstable angina pectoris.
* History of myocardial infarction, stroke, electrocardiographic ischaemia (except stable angina), or life-threatening arrhythmia within the prior 6 months.
* Atrial tachyarrhythmia (eg. atrial fibrillation/flutter) with a heart rate of >100 beats per minute at screening.
* Child-Pugh class B liver disease or liver function abnormalities.
* Clinically significant chronic haematological disease or bleeding disorder
* History of significant peptic ulcer disease within one year before Visit 1
* Resting hypotension (a resting systolic blood pressure of <90 mm Hg) or hypertension (a resting systolic blood pressure >170 mm Hg or a resting diastolic blood pressure >110 mm Hg).
* Symptomatic postural hypotension within the six months of Visit 1.
* Uncontrolled diabetes mellitus (haemoglobin A1c > 12%).
* Patients who are taking nitrates or nitric oxide donors (e.g. molsidomine).
* Patients who are taking anticoagulants, with the exception of anti-platelet agents.
* Patients who are taking androgens (e.g. testosterone), trazodone or anti-androgens.
* Patients who are taking the following inhibitors of cytochrome P 450 CYP 3A4: potent HIV protease inhibitors (ritonavir, indinavir), the anti-mycotic agents itraconazole and ketoconazole (topical forms are allowed) or erythromycin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2003-04; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy comparison is EF domain of the IIEF, vardenafil preferred dose versus placebo at week 18 (after 4 weeks of preferred treatment). | At week 18 (after 4 weeks of preferred treatment).

SECONDARY OUTCOMES:
The relationship between the change from baseline score for; EF domain, SEP2, SEP3 and GEQ with that for ED-QoL and EDITS will be explored for the vardenafil 10mg and 20mg groups respectively | Baseline and at week 18 (after 4 weeks of preferred treatment).
Global Assessment Question (GAQ) responses | At weeks 4, 8, 12, 18 and 26
Treatment groups will be compared with respect to the incidence rates of premature termination, adverse events, lab abnormalities, ECG abnormalities, and concomitant medication use | Baseline and at weeks 4, 8, 12, 18 and 26
Measurements and changes from baseline in vital signs (blood pressure and pulse rate), continuous laboratory variables, ECG cardiac cycle measurements, and ECG heart rate | Baseline and Week 26
Measurements and changes from baseline in vital signs (blood pressure and pulse rate), continuous laboratory variables, | Baseline and at weeks 4, 8, 12, 18 and 26

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- Dublin, Dublin, Ireland
- United Kingdom (21):
  - Reading, Berkshire
  - Durham, County Durham
  - Rhyl, Denbighshire
  - Plymouth, Devon
  - Dublin, Dublin
  - London, Greater London
  - Manchester, Greater Manchester
  - Portsmouth, Hampshire
  - Northwood, Middlesex
  - Norwich, Norfolk
  - Belfast, Northern Ireland
  - Chipping Norton, Oxfordshire
  - Shrewsbury, Shropshire
  - Cardiff, South Glamorgan
  - Doncaster, South Yorkshire
  - Lichfield, Staffordshire
  - Glasgow, Strathclyde
  - Hamilton, Strathclyde
  - Motherwell, Strathclyde
  - Coventry, Warwickshire
  - Leeds, West Yorkshire